CLINICAL TRIAL: NCT00952757
Title: Changes in Hyperprolactinemia Secondary to Antipsychotics After Switching to Quetiapine: a Naturalistic, Prospective, Multicentric Observational Study of 6 Months Follow-up
Brief Title: Changes in Hyperprolactinemia Secondary to Antipsychotics After Switching to Quetiapine
Status: Completed | Type: Observational
Sponsor: Investigaciones Médicas Montejo S.L. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Angel Luis Montejo Gonzalez, University of Salamanca. Hospital Universitario Salamanca. Spain
Other Study IDs: D1443L00008; ANG-QUE-2006-1
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: APS-related Hyperprolactinaemia; Schizophrenia; Bipolar Disorder
Keywords: APS-related hyperprolactinaemia; Quetiapine; Schizophrenia; Bipolar
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1.: Patients diagnosed of schizophrenia or bipolar disorder with APS-related hyperprolactinaemia who have been switched to quetiapine based on the clinician's judgement

SUMMARY:
Hyperprolactinaemia is a common side effect of some antipsychotics (APS), including some atypicals. Clinical consequences of hyperprolactinaemia are broad including amenorrhea, galactorrhea, tender breasts, gynecomastia and sexual dysfunction. Less known but also present is the increased cardiovascular risk, specially in women, disorders of osteoporotic type and a potential increased risk of breast and prostate cancer.

Despite this growing evidence, there are no consistent published data in order to adopt evidence-based decisions that may be beneficial for the patient.

This naturalistic observational 6 months follow-up study on patients with APS-induced hyperprolactinemia aims to obtain more information about the switching approach in cases of hyperprolactinemia secondary to APS and to better establish the role of switching to quetiapine (APS not related with the increase prolactin levels) in this problem.

DETAILED DESCRIPTION:
Hyperprolactinaemia is a common side effect of some antipsychotics (APS), including some atypicals. Clinical consequences of hyperprolactinaemia include most remarkably the appearance of amenorrhea, galactorrhea, tender breasts, and gynecomastia - associated with dysmorphophobia and psychological disorders in some cases, particularly in men-. Another common side effect is sexual dysfunction, with decreased libido, anorgasmia, and in men, impotence, reduced volume ejaculated and even backward ejaculation. Less known but also present is the increased cardiovascular risk, specially in women, disorders of osteoporotic type. Furthermore, several authors have related hyperprolactinemic states with the development of breast cancer including a potential worse prognosis of it (Mandala, 1999; Clevenger 2003; Mujagic, 2004), and with the development of metastatic prostate cancer and resistance to hormone therapy in men (Lisonni, 2005)

Despite this growing evidence and the fact that APS with no apparent increase of prolactin levels exist, such as quetiapine or aripiprazole, many clinicians don't even monitor prolactin levels in patients following APS treatment. And when they do, they find there are no consistent published data in order to adopt evidence-based decisions that may be beneficial for the patient.

This naturalistic observational 6 months follow-up study on patients with APS-induced hyperprolactinemia aims to obtain more information about the switching approach in cases of hyperprolactinemia secondary to APS and to better establish the role of switching to quetiapine in this problem.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature.
* Men aged 18-50 years and women aged 18-45 years.
* Patients diagnosed of schizophrenia or bipolar disorder according to DSM-IV and on ambulatory psychiatric follow-up.
* Treated with one or more antipsychotics other than quetiapine for at least 8 weeks prior to inclusion in the study.
* Prolactin serum levels over 20 ug/L.
* That, in the opinion of the clinician, the origin of the hyperprolactinemia is the antipsychotic treatment administered previously to the patient.
* Switching from previous antipsychotic treatment to quetiapine following the clinical criterion of the investigator in response to hyperprolactinemia in a period less than 5 days prior to inclusion in the study.
* Women with child-bearing potential using an effective contraceptive method and with a negative result in the pregnancy HCG test at the time of inclusion.
* Be able to understand and meet the study requirements.

Exclusion Criteria:

* Pregnant or nursing women.
* Mental retardation.
* Dependence or abuse of substances on inclusion according to DSM-IV criteria.
* Patients that, in the investigator's opinion, are at a high risk of suicide or mean a risk of aggression to others.
* Treated with any of the following drugs that can modify PRL levels on inclusion and during the study: antipsychotics, except for quetiapine, antidepressants -except for mirtazapine-, hormone therapy, spermicides, antiparkinson drugs or dopaminergic agonists, metoclopramide, domperidone, cimetidine or ranitidine, verapamil, enalapril, alpha-methyldopa, reserpine, morphine and other opioid derivatives, anti-retrovirals (protease inhibitors), vitamin D or any complex containing it. These drugs are excluded for their known potential effect on prolactin serum levels, sexual hormones and/or cortisol.
* Administration of an antipsychotic depot injection in one of the usual administration intervals of the depot (e.g., 3-4 weeks) prior to inclusion.
* Be treated with any of the following P450-3A4 cytochrome inhibitors in the 14 days prior to inclusion, including: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, fluvoxamine, indinavir, nelfinavir, ritonavir and saquinavir.
* Be treated with any of the following P450-3A4 cytochrome inducers in the 14 days prior to inclusion, including: phenytoin, carbamazepine, barbiturates, rifampicin, St. John's wart, and glucocorticoids.
* Any contraindication to the use of quetiapine fumarate in the investigator's opinion (including lack of response to it in previous treatment attempts) (applies also to any other treatment to be used in the study -comparative agents-).
* Suffer any medical condition that can effect the absorption, distribution, metabolism or excretion of the study treatment(s).
* Suffer any medical condition in decompensation or not receiving inappropriate treatment for it in the investigator's opinion (e.g., diabetes, angina pectoris, hypertension...) and can affect psychotic symptoms and/or levels of prolactin, sexual hormones and/or cortisol.
* Suffering unstable diabetes.
* Absolute neutrophil count £1.5 x 109 per litre.
* Non-compliance with the study plan.
* Participation in a clinical trial in the four weeks prior to inclusion in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients diagnosed with schizophrenia or bipolar disorder who developed APS-related hyperprolactinaemia and were switched to quetiapine based on the clinician's judgement
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Variation in prolactin serum levels after switching to quetiapine | From baseline to endpoint (month 6)

SECONDARY OUTCOMES:
Changes in the clinical symptoms related to hyperprolactinemia | Baseline to endpoint (month 6)

CONTACTS AND LOCATIONS:
Overall Officials: Ángel L Montejo, Dr, Study Chair — University of Salamanca
Locations (6):
- Spain (6):
  - Servicio de Psiquiatría, Ávila
  - Servicio de Psiquiatria, Burgos
  - Hospital San Telmo, Palencia
  - Hospital Universitario de Salamanca, Salamanca
  - Servicio de Psiquiatria de Valladolid, Valladolid
  - Servicio de Psiquiatría, Zamora